CLINICAL TRIAL: NCT05942651
Title: Reduction of Impulsivity in Patients With Borderline Personality Disorder Using Dual-site Transcranial Magnetic Stimulation
Brief Title: Impulsivity With Borderline Personality Disorder/tMS
Acronym: IMPULSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-A00772-43
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-06

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; brain stimulation; impulsivity
MeSH Terms: conditions — Borderline Personality Disorder; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, parallel-group controlled trial with two arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be block randomized (1:1) to receive either active ccPAS4-ms or sham ccPAS100-ms. Computer generated random numbers will be used to generate the allocation sequence. The allocation sequence will be handled by an independent person from the Administrative Department of the Hospital and will be unavailable to those who enroll and assign patients. Patients will be blind to their treatment assignment. Moreover, the medical doctors who will administer the clinical scales and the researchers that will analyze the data will be blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active ccPAS4-ms (Active Comparator): Device: Magstim BiStim 2002 (The Magstim Company Ltd., Spring Gardens, Whitland, UK) and two small coils (40mm, figure-of-eight coils, Alpha B.I).
  Coil 1 was positioned over right IFC at a 20° angle to the coronal plane with the handle pointing anteriorly, and coil 2 was positioned over right pre- SMA perpendicular to the midline.
  The first stimulation will be applied to the IFC and the second to the pre-SMA, with an interstimulation interval set at 4 ms. A total of 180 stimulation pairs will be delivered every 2 s. (5Hz) for a total duration of 15 minutes at an intensity of 120% of rMT
  Interventions: Device: Non-invasive brain stimulation protocol (Cortico-cortical paired associative stimulation protocol (ccPAS)) delivered at 4 ms intervals.
- Control condition ccPAS100-ms. (Sham Comparator): Device: Magstim BiStim 2002 (The Magstim Company Ltd., Spring Gardens, Whitland, UK) and two small coils (40mm, figure-of-eight coils, Alpha B.I).
  Coil 1 was positioned over right IFC at a 20° angle to the coronal plane with the handle pointing anteriorly, and coil 2 was positioned over right pre- SMA perpendicular to the midline.
  The first stimulation will be applied to the IFC and the second to the pre-SMA, with an interstimulation interval set at 100 ms. A total of 180 stimulation pairs will be delivered every 2 s. (5Hz) for a total duration of 15 minutes at an intensity of 120% of rMT
  Interventions: Device: Non-invasive brain stimulation protocol (Cortico-cortical paired associative stimulation protocol (ccPAS)) delivered at 100 ms intervals

INTERVENTIONS:
Device: Non-invasive brain stimulation protocol (Cortico-cortical paired associative stimulation protocol (ccPAS)) delivered at 4 ms intervals. — The first stimulation will be applied to the IFC and the second to the pre-SMA, with an interstimulation interval set at 4 ms. A total of 180 stimulation pairs will be delivered every 2 s. (5Hz) for a total duration of 15 minutes at an intensity of 120% of rMT
  Arms: active ccPAS4-ms
Device: Non-invasive brain stimulation protocol (Cortico-cortical paired associative stimulation protocol (ccPAS)) delivered at 100 ms intervals — The first stimulation will be applied to the IFC and the second to the pre-SMA, with an interstimulation interval set at 100 ms. A total of 180 stimulation pairs will be delivered every 2 s. (5Hz) for a total duration of 15 minutes at an intensity of 120% of rMT
  Arms: Control condition ccPAS100-ms.

SUMMARY:
This is a prospective, randomized, double-blind, parallel-group controlled trial. The aim of this research project is to compare the clinical benefits achieved in patients with Borderline Personality Disorder (BPD) following two types of intervention: ccPAS active or ccPAS sham.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a mental disorder characterized by unstable interpersonal relationships, emotional lability and marked impulsivity. The latter manifests itself through risky behaviors such as substance abuse, self-harm and suicidal behavior.

Studies suggest that 1.3% of the general population suffers from BPD. However, in clinical settings, BPD patients represent 20% of all inpatients in psychiatric wards and up to 50% of patients hospitalized in emergency departments following a suicide attempt (SA). Moreover, it is estimated that nearly 84% of BPD patients will make at least one SA in their lifetime and up to 10% of them will die by suicide, a rate 50 times higher than the general population. Impulsivity, reflected in difficulties holding back action or stopping an action that has already begun, is one of the key symptoms of BPD.

Recent advances in non-invasive brain stimulation have led to the emergence of a new stimulation protocol known as Paired Cortico-Cortical Associative Stimulation (ccPAS), which consists of repeating paired stimulations using two TMS coils placed respectively on two cortical regions of interest. Paired stimulations' repetition induces plasticity by strengthening synaptic connectivity between the two targeted regions.

The aim of this project is to test the efficacy of a ccPAS protocol in enhancing effective connectivity between the IFC and pre-SMA in order to reduce impulsivity in BPD patients.

The Sponsor hypothesized that one ccPAS session, using two coils simultaneously, targeting the IFC and pre-SMA with a 'physiological' inter-stimulus interval of 4ms will improve motor inhibition abilities (reduce SSRT), compared to the group receiving 'control' ccPAS (100ms inter-stimulus interval (ccPAS100-ms)).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD (established by a psychiatrist and confirmed in a structured interview using the MINI) based on the Diagnostic and Statistical Manual of Mental Disorders (DSM V).

Exclusion Criteria:

* Contraindications to TMS/MRI (pacemakers or other devices likely to interfere with the magnetic field).
* Pregnant or breast-feeding women.
* Ongoing anxiolytic treatment (benzodiazepines), neuroleptic treatment or anticonvulsants acting on GABAergic transmission ; 24 hours prior to the protocol.
* Diagnosis of other chronic psychiatric pathology including bipolar disorder type I or II and addictions (except tobacco).
* Protective measure (curatorship or guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Significant reduction in reaction time of the Emotional Stop Signal (SSRT) for the ccPAS4-ms group compared to the ccPAS100-ms sham group | 2 times: Outcome measure will be assessed: immediately before the ccPAS protocol and immediately after the ccPAS protocol, for both groups
  The ability to inhibit an action (motor inhibition) is quantified using a 'Stop Signal' task in which the reaction time required to inhibit the action (SSRT) is calculated. The longer the SSRT, the poorer the ability to inhibit an action and the greater the motor impulsivity

SECONDARY OUTCOMES:
Increased effective inhibitory connectivity within the fronto-striatal network (DLPFC-M1), intracortical inhibition (short and long interval) and cortical silent period for the ccPAS4-ms group, when compared with the ccPAS100-ms group | 2 times: Outcome measure will be assessed: immediately before the ccPAS protocol and immediately after the ccPAS protocol, for both groups
  Dual-site transcranial magnetic stimulation (TMS) can be used to probe effective connectivity between the left DLPFC and the left M1 (Wang et al. 2021). Conditioned motor evoked potential (MEP) amplitude evoked by dual-site TMS and measured with surface electromyography (EMG) is compared to MEP amplitude evoked by TMS applied over M1 alone.
Levels of intracortical inhibition within M1. | 1 time: Measured before the ccPAS protocol, in both groups.
  Paired-pulse TMS provides a non-invasive method to study intracortical inhibitory circuits. Short-interval intracortical inhibition (SICI) is a well-established paired-pulse measure of inhibitory circuitry within the M1 area. SICI results from a subthreshold conditioning stimulus (CS) followed 3.5 ms later by a suprathreshold test stimulus (TS) delivered through the same coil over M1. This measurement will be correlated with the other inhibition measurements (SSRT at baseline and duration of the silent period) to provide an overall view of the efficacy/inefficacy of this inhibitory system in patients with borderline personality disorder.
Duration of cortical silence period (in ms). | 1 time: Measured before the ccPAS protocol, in both groups
  Single-pulse TMS applied over M1 during a voluntary contraction elicited a motor evoked potential followed immediately by a period of EMG silence that has been assumed to reflect intracortical inhibition. This measurement will be correlated with the other inhibition measurements (SSRT at baseline and SICI) to provide an overall view of the efficacy/inefficacy of this inhibitory system in patients with borderline personality disorder.
Cognitive task manipulating environment-emotion-behavior interactions. | 1 time: Measured before the ccPAS protocol, in both groups.
  The task is framed to participants as being a fish gathering algae while predators might approach for which they need to check and if appropriate hide. The task features differentially evoke emotions of stress and excitement. Self-reported stress and threat-avoidance behaviors during the task will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, AURA, France

IPD SHARING:
Plan to Share IPD: No